CLINICAL TRIAL: NCT00570973
Title: A Randomized, Controlled, Multicentric Trial Comparing Endoscopic Band Ligation Versus Ransjugular Intrahepatic Portosystemic Stent Shunt in Cirrhotic Patients With Recurrent Variceal Bleeding Non Responding to Medical Therapy
Brief Title: Band Ligation Versus Transjugular Intrahepatic Portosystemic Stent Shunt (TIPS) in Cirrhotics With Recurrent Variceal Bleeding Non Responding to Medical Therapy
Acronym: ENDOvsTIPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Arnulf Ferlitsch, MD, Gastroenterology and Hepatology, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ENDOvsTIPS
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Gastrointestinal Hemorrhage; Variceal Bleeding; Cirrhosis; Encephalopathy
Keywords: Variceal Bleeding; Cirrhosis; Encephalopathy; Endoscopic band ligation; TIPS
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Fibrosis; Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Endoscopic Band ligation combined with medical therapy (orally, daily administered propranolol and mononitrate)
  Interventions: Procedure: endoscopic band ligation
- 2 (Active Comparator): Transjugular intrahepatic portosystemic stent shunt with PTFE-covered stent
  Interventions: Procedure: TIPS-Implantation

INTERVENTIONS:
Procedure: endoscopic band ligation — Endoscopic Band ligation of esophageal varices, performed every 2-4 weeks until resolution of varices
  Arms: 1
Procedure: TIPS-Implantation — Transjugular intrahepatic portosystemic stent shunt with PTFE-covered stent, placed once, under fluoroscopic control,
  Arms: 2

SUMMARY:
Patients with liver cirrhoses and recent history of variceal bleeding, with HVPG documented non response to medical therapy with non selective beta blockers +/- mononitrates or variceal rebleeding during adequate medical therapy will be randomized to undergo either multi-session endoscopic multi-band ligation and continuation of medication or TIPS placement. Best treatment for this group of cirrhotic patients is not known so far.

DETAILED DESCRIPTION:
Reduction of portal pressure are with oral intake of non selective beta blockers, often combined with mononitrates are the method of choice in secondary prophylaxis of esophageal variceal bleeding. However, studies have shown that this therapy is effective only in 20-50% of the patients, documented by a significant drop of the portal pressure with hepatic venous pressure (HVPG) measurements. The best method for secondary prevention in this high risk patient cohort is not known so far. In this randomized controlled study we hypothesise, that a group of 20 vs 20 patients is large enough to discriminate efficacy of prevention of rebleeding in patients receiving TIPS implantation or endoscopic band ligation in patients non responding to medical therapy as secondary prophylaxis of esophageal variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis
* bleeding from esophageal varices within the last 6 months
* sufficient medical therapy (at least 80 mg propranolol per day)
* signed written informed consent

Exclusion Criteria:

* bleeding of gastric varices
* portal vein thrombosis
* insufficient medical therapy (less than 80 mg propranolol per day)
* exclusion criteria for TIPS/band ligation (anatomy, impaired coagulation parameters, severe encephalopathy, severe liver failure (bilirubin > 10 mg/dl)) congestive heart failure, pulmonary hypertension, polycystic liver disease, presence or suspicion of active systemic, biliary or ascitic fluid infection, known cavernous portal vein occlusion
* Budd Chiari syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Recurrence of Variceal Bleeding | 2 years

SECONDARY OUTCOMES:
Survival of Patients | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Ferlitsch, MD, Principal Investigator — Medical University of Vienna
Locations (4):
- Austria (4):
  - Internal Medicine IV, Krankenhaus der Elisabethinen Linz, Linz, Upper Austria
  - Medical University of Graz, Graz
  - Dept. of Internal Medicine III, Gastroenterology and Hepatology, Medical University of Vienna, Vienna
  - Wilhelminenspital der Stadt Wien, Vienna

REFERENCES:
- [Derived] Simonetti RG, Perricone G, Robbins HL, Battula NR, Weickert MO, Sutton R, Khan S. Portosystemic shunts versus endoscopic intervention with or without medical treatment for prevention of rebleeding in people with cirrhosis. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD000553. doi: 10.1002/14651858.CD000553.pub3. PMID 33089892